CLINICAL TRIAL: NCT03141450
Title: Plasma Concentrations of Prophylactic Cefazolin in Pediatric Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Plasma Concentrations of Prophylactic Cefazolin in Pediatric Patients Undergoing Cardiac Surgery With CPB
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Saowaphak Lapmahapaisan, Asst. Prof., Mahidol University
Other Study IDs: 449/2559
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgical site infection (SSI) is a serious operative complication that may be associated with any surgical procedures. It increases morbidity and mortality after cardiac surgery. Plasma concentration of prophylactic antibiotic, routinely cefazolin, is altered by effects of cardiopulmonary bypass. This study is conducted to measure the plasma concentrations of cefazolin to determine its adequacy in pediatric patients undergoing elective cardiac surgery with cardiopulmonary bypass including its correlation with the incidence of postoperative SSI.

ELIGIBILITY:
Inclusion Criteria:

1. age < 7 years old
2. undergoing elective cardiac surgery with cardiopulmonary bypass
3. receive cefazolin as prophylactic antibiotic

Exclusion Criteria:

1. Known or family history of penicillin or cephalosporins allergy
2. Coexisting liver or renal disease
3. Previous infection or received any antibiotics within 4 weeks
4. Previous surgery with median sternotomy
5. Predicted cardiopulmonary bypass time of less than 30 minutes or more than 150 minutes
6. Severe hemodynamic instability during the operation, requiring mechanical circulatory support

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients whose age less than 7 years old, undergo elective cardiac surgery with cardiopulmonary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
plasma concentration of cefazolin in pediatric cardiopulmonary bypass | 12 hours
  plasma concentration of cefazolin

SECONDARY OUTCOMES:
incidence of surgical site infection after elective pediatric cardiac surgery | 30 days
  surgical site infection

CONTACTS AND LOCATIONS:
Overall Officials: Saowaphak Lapmahapaisan, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Thailand